CLINICAL TRIAL: NCT02407327
Title: Trattamento Personalizzato Del Tumore NSCLC Avanzato: Potenziali Applicazioni Della Caratterizzazione Fenotipica e Molecolare Delle Cellule Tumorali Circolanti (CTC)
Brief Title: Individualized Treatment of Patients With Advanced NSCLC: Potential Application for Circulating Tumor Cells (CTC) Molecular and Phenotypical Profiling
Acronym: 2012/52
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: GR-2010-2303193
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Circulating tumour cells in Advanced Non Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the percentage of CTC-positive patients and total CTC numbers in patients with advanced Non Small Cell Lung Cancer .

DETAILED DESCRIPTION:
The primary aim of the Project is to determine the percentage of CTC-positive patients and total CTC numbers in advanced NSCLC at baseline, before starting treatment.

To valuate CTC count modifications as an early predictor of response to treatment a prospective observational study will be conducted, consecutively enrolling 150 patients regardless of type or line of therapy, which will be reevaluated for disease status and CTC count depending on the type and schedule of treatment.

Furthermore, purified CTC will be obtained by automated platform and DNA sequencing will be performed to assess sensitizing mutations in advanced NSCLC patients. The EGFR mutations or EML4-ALK fusion gene detected in CTC will be compared with those reported for the tumor specimen using standard sequencing.

In parallel, the CTC count assay will be integrated with mAb targeting EGFR or EML4-ALK fusion gene, to test whether assaying the quote of EGFR-positive and ALK-positive CTC provides a more sensitive marker for rating pharmacodynamic effects in patients compared with total CTC counts.

Moreover, it was reported that NSCLC cells with EGFR mutations manifest activation of the PI3K (phosphatidylinositol 3-kinase)-AKT and MEK-ERK (extracellular signal-regulated kinase) signaling pathways under the control of EGFR, and exposure of such cells to EGFR-TKIs blocks signaling by both pathways and induces apoptosis 13. To evaluate whether live vs. apoptotic CTC changes under treatment may be used as predictor of tumor response, M30-positive CTC will be quantified as previously 8.

Data obtained with the CTC assay will be correlated with common prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, males or females;
* Patients with NSCLC confirmed by histopathology or cytology;
* Life expectancy > 6 months;
* Patients are voluntary to participate and sign the informed contents

Exclusion Criteria:

* Any condition which might hamper compliance to the schedule of assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change of CTC count during treatment and comparison with CT and PET | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, PD, Italy

REFERENCES:
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Mitsudomi T, Morita S, Yatabe Y, Negoro S, Okamoto I, Tsurutani J, Seto T, Satouchi M, Tada H, Hirashima T, Asami K, Katakami N, Takada M, Yoshioka H, Shibata K, Kudoh S, Shimizu E, Saito H, Toyooka S, Nakagawa K, Fukuoka M; West Japan Oncology Group. Gefitinib versus cisplatin plus docetaxel in patients with non-small-cell lung cancer harbouring mutations of the epidermal growth factor receptor (WJTOG3405): an open label, randomised phase 3 trial. Lancet Oncol. 2010 Feb;11(2):121-8. doi: 10.1016/S1470-2045(09)70364-X. Epub 2009 Dec 18. PMID 20022809
- [Background] Amadori A, Rossi E, Zamarchi R, Carli P, Pastorelli D, Jirillo A. Circulating and disseminated tumor cells in the clinical management of breast cancer patients: unanswered questions. Oncology. 2009;76(6):375-86. doi: 10.1159/000215581. Epub 2009 Apr 30. PMID 19407470
- [Background] Meng S, Tripathy D, Shete S, Ashfaq R, Haley B, Perkins S, Beitsch P, Khan A, Euhus D, Osborne C, Frenkel E, Hoover S, Leitch M, Clifford E, Vitetta E, Morrison L, Herlyn D, Terstappen LW, Fleming T, Fehm T, Tucker T, Lane N, Wang J, Uhr J. HER-2 gene amplification can be acquired as breast cancer progresses. Proc Natl Acad Sci U S A. 2004 Jun 22;101(25):9393-8. doi: 10.1073/pnas.0402993101. Epub 2004 Jun 11. PMID 15194824
- [Background] de Bono JS, Attard G, Adjei A, Pollak MN, Fong PC, Haluska P, Roberts L, Melvin C, Repollet M, Chianese D, Connely M, Terstappen LW, Gualberto A. Potential applications for circulating tumor cells expressing the insulin-like growth factor-I receptor. Clin Cancer Res. 2007 Jun 15;13(12):3611-6. doi: 10.1158/1078-0432.CCR-07-0268. PMID 17575225
- [Background] Wang LH, Pfister TD, Parchment RE, Kummar S, Rubinstein L, Evrard YA, Gutierrez ME, Murgo AJ, Tomaszewski JE, Doroshow JH, Kinders RJ. Monitoring drug-induced gammaH2AX as a pharmacodynamic biomarker in individual circulating tumor cells. Clin Cancer Res. 2010 Feb 1;16(3):1073-84. doi: 10.1158/1078-0432.CCR-09-2799. Epub 2010 Jan 26. PMID 20103672
- [Background] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Background] Hofman V, Ilie MI, Long E, Selva E, Bonnetaud C, Molina T, Venissac N, Mouroux J, Vielh P, Hofman P. Detection of circulating tumor cells as a prognostic factor in patients undergoing radical surgery for non-small-cell lung carcinoma: comparison of the efficacy of the CellSearch Assay and the isolation by size of epithelial tumor cell method. Int J Cancer. 2011 Oct 1;129(7):1651-60. doi: 10.1002/ijc.25819. Epub 2011 Mar 11. PMID 21128227
- [Background] Krebs MG, Sloane R, Priest L, Lancashire L, Hou JM, Greystoke A, Ward TH, Ferraldeschi R, Hughes A, Clack G, Ranson M, Dive C, Blackhall FH. Evaluation and prognostic significance of circulating tumor cells in patients with non-small-cell lung cancer. J Clin Oncol. 2011 Apr 20;29(12):1556-63. doi: 10.1200/JCO.2010.28.7045. Epub 2011 Mar 21. PMID 21422424
- [Background] Sakairi Y, Nakajima T, Yasufuku K, Ikebe D, Kageyama H, Soda M, Takeuchi K, Itami M, Iizasa T, Yoshino I, Mano H, Kimura H. EML4-ALK fusion gene assessment using metastatic lymph node samples obtained by endobronchial ultrasound-guided transbronchial needle aspiration. Clin Cancer Res. 2010 Oct 15;16(20):4938-45. doi: 10.1158/1078-0432.CCR-10-0099. Epub 2010 Oct 5. PMID 20926401
- [Background] Tracy S, Mukohara T, Hansen M, Meyerson M, Johnson BE, Janne PA. Gefitinib induces apoptosis in the EGFRL858R non-small-cell lung cancer cell line H3255. Cancer Res. 2004 Oct 15;64(20):7241-4. doi: 10.1158/0008-5472.CAN-04-1905. PMID 15492241
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Pirker R, Herth FJ, Kerr KM, Filipits M, Taron M, Gandara D, Hirsch FR, Grunenwald D, Popper H, Smit E, Dietel M, Marchetti A, Manegold C, Schirmacher P, Thomas M, Rosell R, Cappuzzo F, Stahel R; European EGFR Workshop Group. Consensus for EGFR mutation testing in non-small cell lung cancer: results from a European workshop. J Thorac Oncol. 2010 Oct;5(10):1706-13. doi: 10.1097/JTO.0b013e3181f1c8de. PMID 20871269
- [Background] Schwarzenbach H, Chun FK, Isbarn H, Huland H, Pantel K. Genomic profiling of cell-free DNA in blood and bone marrow of prostate cancer patients. J Cancer Res Clin Oncol. 2011 May;137(5):811-9. doi: 10.1007/s00432-010-0941-5. Epub 2010 Aug 4. PMID 20683729
- [Background] Amadori A, Zamarchi R, De Silvestro G, Forza G, Cavatton G, Danieli GA, Clementi M, Chieco-Bianchi L. Genetic control of the CD4/CD8 T-cell ratio in humans. Nat Med. 1995 Dec;1(12):1279-83. doi: 10.1038/nm1295-1279. PMID 7489409
- [Background] Rossi E, Fassan M, Aieta M, Zilio F, Celadin R, Borin M, Grassi A, Troiani L, Basso U, Barile C, Sava T, Lanza C, Miatello L, Jirillo A, Rugge M, Indraccolo S, Cristofanilli M, Amadori A, Zamarchi R. Dynamic changes of live/apoptotic circulating tumour cells as predictive marker of response to sunitinib in metastatic renal cancer. Br J Cancer. 2012 Oct 9;107(8):1286-94. doi: 10.1038/bjc.2012.388. Epub 2012 Sep 6. PMID 22955853
- [Background] de Haas EC, di Pietro A, Simpson KL, Meijer C, Suurmeijer AJ, Lancashire LJ, Cummings J, de Jong S, de Vries EG, Dive C, Gietema JA. Clinical evaluation of M30 and M65 ELISA cell death assays as circulating biomarkers in a drug-sensitive tumor, testicular cancer. Neoplasia. 2008 Oct;10(10):1041-8. doi: 10.1593/neo.08620. PMID 18813353
- [Background] Punnoose EA, Atwal SK, Spoerke JM, Savage H, Pandita A, Yeh RF, Pirzkall A, Fine BM, Amler LC, Chen DS, Lackner MR. Molecular biomarker analyses using circulating tumor cells. PLoS One. 2010 Sep 8;5(9):e12517. doi: 10.1371/journal.pone.0012517. PMID 20838621
- [Background] PubMed ID:17575225
- [Background] Rossi E, Basso U, Celadin R, Zilio F, Pucciarelli S, Aieta M, Barile C, Sava T, Bonciarelli G, Tumolo S, Ghiotto C, Magro C, Jirillo A, Indraccolo S, Amadori A, Zamarchi R. M30 neoepitope expression in epithelial cancer: quantification of apoptosis in circulating tumor cells by CellSearch analysis. Clin Cancer Res. 2010 Nov 1;16(21):5233-43. doi: 10.1158/1078-0432.CCR-10-1449. Epub 2010 Oct 26. PMID 20978147